CLINICAL TRIAL: NCT06490354
Title: Effectiveness of the Use of Lightback in Conventional Football Training. Randomised Clinical Trial.
Brief Title: Effectiveness of the Use of Lightback in Conventional Football Training.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 290624
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Injury; Hip
Keywords: hip; gluteal regions; range of motion, articular; footballs
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lightback group (Experimental): Use of the lightback device to relax the gluteal musculature.
  Interventions: Device: Lightback group
- Conventional group (Active Comparator): Conventional treatment to relax the gluteal musculature and prevent hamstring injuries.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Device: Lightback group — Use of the patented Lightback device to relax the gluteal musculature and prevent hamstring injuries.
  Arms: Lightback group
Other: Conventional treatment — Conventional treatment to relax the gluteal musculature and prevent hamstring injuries.
  Arms: Conventional group

SUMMARY:
Lightback is a patented device that allows instrumental stretching of the gluteal muscles. Football players overload this musculature and this type of device is effective and the cost/benefit ratio is high.

The intention is to carry out a randomised clinical trial to carry out a study on athletes to see the differences between a group of football players with their normal training and a group of football players with their normal training and the application of lightback beforehand.

The variables studied will be sprint speed in 20 and 40m, vertical jump height, hamstring muscle injuries throughout the season, triceps sural injuries throughout the season, internal and external hip ROM, dorsal flexion ankle ROM.

ELIGIBILITY:
Inclusion Criteria:

* Professional football players
* Age range 18 to 45 years
* Able to perform physical exertion without discomfort.

Exclusion Criteria:

* Football players recently injured or in an active recovery phase.
* Heterometrics
* Non-collaborators
* Alteration of sensitivity

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Range of motion | 5 weeks
  Measurement of hip joint range and ankle dorsiflexion measured with goniometer

SECONDARY OUTCOMES:
Sprint | 5 weeks
  Measurement of speed over 20 and 40 metres using approved devices
Vertical jump height | 5 weeks
  Measurement of height (metres) using approved devices

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fernandes CA, Norte GE, Schwab SM, Gokeler A, Murray A, Bazett-Jones DM, Sherman DA. Interpersonal Coordination between Female Soccer Players: Leader-Follower Roles within a Collision-Avoidance Task. Int J Sports Phys Ther. 2024 May 1;19(5):548-560. doi: 10.26603/001c.116156. eCollection 2024. PMID 38707861
- [Result] Junge A, Dvorak J. Soccer injuries: a review on incidence and prevention. Sports Med. 2004;34(13):929-38. doi: 10.2165/00007256-200434130-00004. PMID 15487905
- [Result] Pirri C, Pirri N, Guidolin D, Macchi V, Porzionato A, De Caro R, Stecco C. Ultrasound Imaging in Football Players with Previous Multiple Ankle Sprains: Keeping a Close Eye on Superior Ankle Retinaculum. Bioengineering (Basel). 2024 Apr 25;11(5):419. doi: 10.3390/bioengineering11050419. PMID 38790287
- [Result] Al Attar WSA, Soomro N, Sinclair PJ, Pappas E, Sanders RH. Effect of Injury Prevention Programs that Include the Nordic Hamstring Exercise on Hamstring Injury Rates in Soccer Players: A Systematic Review and Meta-Analysis. Sports Med. 2017 May;47(5):907-916. doi: 10.1007/s40279-016-0638-2. PMID 27752982
- [Result] Biz C, Nicoletti P, Baldin G, Bragazzi NL, Crimi A, Ruggieri P. Hamstring Strain Injury (HSI) Prevention in Professional and Semi-Professional Football Teams: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Aug 4;18(16):8272. doi: 10.3390/ijerph18168272. PMID 34444026
- [Result] Petersen J, Thorborg K, Nielsen MB, Budtz-Jorgensen E, Holmich P. Preventive effect of eccentric training on acute hamstring injuries in men's soccer: a cluster-randomized controlled trial. Am J Sports Med. 2011 Nov;39(11):2296-303. doi: 10.1177/0363546511419277. Epub 2011 Aug 8. PMID 21825112
- [Result] Lovell R, Knox M, Weston M, Siegler JC, Brennan S, Marshall PWM. Hamstring injury prevention in soccer: Before or after training? Scand J Med Sci Sports. 2018 Feb;28(2):658-666. doi: 10.1111/sms.12925. Epub 2017 Jun 28. PMID 28544170